CLINICAL TRIAL: NCT05137808
Title: A Prospective Cohort Study, Understanding Blood Pressure Changes in the Immediate Twelve Weeks Postpartum for Women Who Had a Hypertensive Disorder in Pregnancy and How Existing Care Pathways Identify and Monitor Women at Risk of Cardiovascular Disease
Brief Title: Understanding Blood Pressure Changes After Birth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021.0199
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Hypertension in Pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Research Question How does maternal blood pressure respond in the postpartum period for women who had a hypertensive disorder in pregnancy?

Aim To evaluate the recovery of maternal blood pressure after a pregnancy affected by new onset hypertension after twenty weeks gestation

Objectives

* To identify rates of persistent hypertension after pregnancies affected by HDP
* To assess and compare the accuracy of HBPM against the gold standard of ABPM
* To assess the maternal acceptance of HBPM and ABPM
* To explore what CVD-related care information is provided at the 6-8 week GP appointment

DETAILED DESCRIPTION:
This research aims to investigate how women's blood pressure responds after birth and assess the time it takes to return to normal ranges. This will be calculated by participants undertaking three consecutive days of home blood pressure monitoring, every fortnight from two until twelve weeks postpartum. At twelve weeks postpartum, women will have a twenty-four ambulatory blood pressure assessment. This will highlight the prevalence of persistent high blood pressure and how often GPs will need to monitor women's blood pressure in the immediate few weeks after birth. Women will be asked to complete a questionnaire after their six to eight week GP appointment, assessing if women recall having their blood pressure checked and/or the risks of heart disease explained to them and if they received any lifestyle advice to reduce these risks. Women will be asked to complete a second questionnaire at twelve weeks postpartum assessing their acceptance and preference of home and twenty four hour blood pressure monitoring. This research aims to identify any gaps in the current care of women in the postnatal period and use this information to provide better quality of care to women so they can lead healthier lives and reduce their risk of heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a confirmed diagnosis of new onset of high blood pressure after twenty weeks gestation
* Maternal Age >16 years old
* Mental capacity to give informed consent
* Ability to be able to communicate to HCP if their BP range is above target (for example women where English is not their first language).

Exclusion Criteria:

• Pre-existing hypertension

Min Age: 16 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be selected via purposive sampling as participants will need to have a diagnosis of gestational hypertension and/or pre-eclampsia to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of persistent hypertension in postpartum period | 12 weeks
  Blood Pressure expressed as mmHg at twelve weeks postpartum via 24 hour ambulatory blood pressure monitoring.

SECONDARY OUTCOMES:
Levels of agreement of diastolic and systolic blood pressures between HBPM and ABPM measurements | 12 weeks
  Accuracy of HBPM for diagnosing hypertension and pre-hypertension will assessed by sensitivity, specificity, PPV and NPV analysis and Cohen's Kappa will measure the agreement between both. ICC and Bland Altman plots will assess agreement between continuous variables (SBP+DBP) and assess for systematic effects.
Identification of women who would benefit from closer BP surveillance | 12 weeks
  Using univariate logistic regression to assess what variables such as age, BMI, ethnicity, etc are associated with persistent hypertension at twelve weeks postpartum.
Key time points when BP should be monitored post birth | 10 weeks
  Based on most prevalent time points when BP is at it's highest according to two weekly intervals from week 2 to week 12 post birth

CONTACTS AND LOCATIONS:
Locations (1):
- St. George's University NHS Hopsitals, Wandsworth, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sheehan E, Wang C, Cauldwell M, Bick D, Thilaganathan B. Understanding maternal postnatal blood pressure changes following hypertensive disorders in pregnancy: protocol for a prospective cohort study. BMJ Open. 2022 Apr 1;12(4):e060087. doi: 10.1136/bmjopen-2021-060087. PMID 35365547